**Document Type:** Informed Consent Form

Official Title: Price Elasticity of Fruit (Shop For Success)

NCT Number: NCT04097262

**IRB Approval Date:** 08/16/2019

# GRAND FORKS HUMAN NUTRITION RESEARCH CENTER CONSENT TO PARTICIPATE IN RESEARCH

**Project Title:** Shop For Success

Principal Investigator: Lisa Jahns, PhD, RD

**Phone/Email Address:** 701-795-8331/lisa.jahns@ars.usda.gov

**Department:** Grand Forks Human Nutrition Research Center (GFHNRC)

#### What should I know about this research?

- Someone will explain this research to you.
- Taking part in this research is voluntary. Whether you take part is up to you.
- If you don't take part, it won't be held against you.
- You can take part now and later drop out, and it won't be held against you.
- If you don't understand, ask questions.
- Ask all the questions you want before you decide.

## How long will I be in this research?

We expect that your taking part in this research will last approximately 1.5 hours.

### Why is this research being done?

The purpose of this research is to study how the price of foods affects food buying choices at the grocery store. We are interested in this topic because the price of foods can have a big impact on what people choose to buy and prices change over time. We are doing this study to see how changes in food prices affect what foods mothers choose for their families.

## What happens to me if I agree to take part in this research?

If you decide to take part in this research study, you will be given play money and asked to "buy" foods in our laboratory-based grocery store. Foods will be symbolized by pictures along with their price. Using your play money, you will be asked to "buy" enough food for your family for a one-week period. During this study we will change the price of certain foods to see how that affects your choice to put them in your grocery cart.

You will be asked to fill out a questionnaire asking about your age, gender, race, ethnicity, income, and people in your household. You will also be asked to fill out questionnaires asking about how you would react to certain money situations, stress, hunger level, and your knowledge about food and health. You are free to skip any questions that you do not prefer to answer. Your height and weight will also be measured.

| Approval Date: | AUG | 16 | 2019 |
|-----------------------|-------|-----|------|
| Expiration Date: | AUG | 15 | 2020 |
| University of North D | akota | IRB | |

| Date: |
|-------------------|
| Subject Initials: |

## Could being in this research hurt me?

The most important risks or discomforts that you may expect from taking part in this research include some awkward feelings answering questions about demographic features and income. It may be possible for some people to be emotionally uncomfortable while answering the questionnaires, but only relevant questions required to determine eligibility and assess factors related to the research will be asked. Any questions or concerns will be addressed by the PI or her delegate.

## Will being in this research benefit me?

It is not expected that you will personally benefit from this research.

Possible benefits to others include that results of this research may give more knowledge about how food price changes affect diet patterns.

## How many people will participate in this research?

Approximately 80 people will take part in this study at the GFHNRC.

#### Will it cost me money to take part in this research?

You will not have any costs for being in this research study. You will be expected to provide your transportation to and from the GFHNRC. We do not withhold income, social security, unemployment taxes, or any other taxes because you are not an employee of the GFHNRC. You may have to pay income taxes on the money you receive. All tax questions relating to the taxability of the payment should be directed to your personal tax accountant or to your local Internal Revenue Service Office. If you are not a United States citizen, check your documentation to make sure you can receive money from a non-University source without risking your status in the United States.

#### Will I be paid for taking part in this research?

You will be paid for being in this research study. You will receive \$70 for being in this research study. You may choose to receive a 2-month individual membership or 2-month family membership to Choice Health & Fitness, instead.

#### Who is funding this research?

The United States Department of Agriculture (USDA) is funding this research study. This means that the GFHNRC is receiving payments from the USDA to support the activities that are required to conduct the study. No one on the research team will receive a direct payment or an increase in salary from the USDA for conducting this study.

### What happens to information collected for this research?

Your private information may be shared with individuals and organizations that conduct or watch over this research, including:

The GFHNRC

| Approval Date: | AUG | 16 | 2019 |
|------------------|-----------|-----|------|
| Expiration Date: | AUG | 15 | 2020 |
| University of No | th Dakota | IRB | |

| Date: |
|-------------------|
| Subject Initials: |

- The USDA, as specified in the USDA/ARS Privacy Act System of Records
- The University of North Dakota (UND) Research Compliance & Ethics Office
- The Institutional Review Board (IRB) that reviewed this research
- Key personnel of this study
- and as required by law or court order.

We may publish the results of this research. However, we will keep your name and other identifying information confidential. We protect your information from disclosure to others to the extent required by law. We cannot promise complete secrecy. Clinical trial information will be submitted to the National Institutes of Health/National Library of Medicine to be included in the clinical trial registry data bank (www.clinicaltrials.gov).

Data or specimens collected in this research might be de-identified and used for future research or distributed to another investigator for future research without your consent.

## What if I agree to be in the research and then change my mind?

If you decide to leave the study early, we ask that you please inform the study coordinator of your decision. Your decision will not affect your current or future relations with the GFHNRC or UND.

## Who can answer my questions about this research?

If you have questions, concerns, or complaints, or think this research has hurt you or made you sick, talk to the research team at the phone number listed above on the first page.

This research is being overseen by an Institutional Review Board ("IRB"). An IRB is a group of people who perform independent review of research studies. You may talk to them at 701.777.4279 or <u>UND.irb@UND.edu</u> if:

- You have questions, concerns, or complaints that are not being answered by the research team.
- You are not getting answers from the research team.
- You cannot reach the research team.
- You want to talk to someone else about the research.
- You have questions about your rights as a research subject.
- You may also visit the UND IRB website for more information about being a research subject: http://und.edu/research/resources/human-subjects/research-participants.html

| Approval Date: | AUG | 1 6 | 2019 |
|---------------------|--------|-------|------|
| Expiration Date: | AUG | 15 | 2020 |
| University of North | Dakota | a IRE | 3 |

| Date: |
|-------------------|
| Subject Initials: |

| if you conse | | | | ou may qual | ify for in the | e future. Please ind | icate |
|---|---|---|---|---|---|---|---|
| (Please circle | e one) | YES | NO | | | | |
| Initials | = | | | | | | |
| Consent:<br>Your signatu<br>form. | ıre docur | nents you | r consent to | take part in | this study. | You will receive a c | юру |
| Subject's Na | ame: | | | | | | |
| Signature of | Subject | | | | | Date | |
| Signature of | Person V | Who Obtai | ined Conser | nt | | Date | |
| Signature of | Person V | Who Obtai | ined Conser | nt | | Date | |
| Signature of | Person V | Who Obtai | ined Conser | nt - | | Date | |
| Signature of | Person V | Who Obtai | ned Conser | nt | | Date | |
| Signature of | Person V | Who Obtai | ined Conser | nt | | Date | |
| Signature of | Person | Who Obtai | ined Conser | nt | | Date | |
| Signature of | | Who Obtai | ned Conser | nt | | Date | |

University of North Dakota IRB

Subject Initials: